CLINICAL TRIAL: NCT04632875
Title: Identifying Neural Correlates of Altruism
Brief Title: Online Trial of Meditation and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-180-2
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2020-11

CONDITIONS: Meditation
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loving-Kindness Meditation (Experimental): 4-week guided Loving-Kindness Meditation training (administered online).
  Interventions: Behavioral: Loving-Kindness Meditation
- Relaxation Meditation (Experimental): 4-week guided Relaxation Meditation training (administered online).
  Interventions: Behavioral: Relaxation Meditation

INTERVENTIONS:
Behavioral: Loving-Kindness Meditation — Approximately 15-minute sessions are administered 6 days per week
  Other Names: Metta Meditation
  Arms: Loving-Kindness Meditation
Behavioral: Relaxation Meditation — Approximately 15-minute sessions are administered 6 days per week
  Other Names: Progressive Muscle Relaxation
  Arms: Relaxation Meditation

SUMMARY:
This study investigates how different types of meditation may affect behaviors and emotions. The study is conducted entirely online and involves listening to 4-weeks of a guided meditation training. The meditation involves either Loving-Kindness or Relaxation techniques. The purpose of the study is to assess changes in behaviors and emotions using standard questionnaires, reports of real-world behavior, and online behavioral tasks. The overarching goal is to help clarify how mind-body practices may improve some aspects of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Is a medically healthy individual
* Lives in the United States
* Has reliable internet access and the ability to join a Zoom video chat

Exclusion Criteria:

* Has experience with meditation or other mind-body practices
* Has a neurological disease
* Has a current psychiatric disorder
* Is on medication that affects the central nervous system (e.g. psychotropic drugs)
* Has recurrent or chronic pain
* Is pregnant or planning to become pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Social functioning | 4-5 weeks
  Participants will complete a questionnaire about their real-world social behaviors. An aggregate score will be computed; higher scores will indicate better social functioning.
Affective responses | 4-5 weeks
  Participants will perform a wall-sit test and responses will be measured using a 0-100 Visual Analog Scale of intensity.

SECONDARY OUTCOMES:
Psychological well-being related to COVID-19 | 4-5 weeks
  Participants will complete a questionnaire related to the psychological impact of COVID-19 social distancing. Higher scores will indicate worse psychological impact of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail A Marsh, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No